CLINICAL TRIAL: NCT07080840
Title: Adherence as a Moderator of Phosphorus Education Effectiveness in Hemodialysis Patients: an Exploratory Study
Brief Title: Phosphorus Education and Adherence in Hemodialysis Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jen-Ai Hospital Institutional Review Board (Industry)
Responsible Party: Principal Investigator, Ming-Chih Chang, Jen-Ai Hospital Principal Investigator, Jen-Ai Hospital Institutional Review Board
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: WHChen
Record Dates: First submitted 2025-06-18; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Nursing Education; Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Nursing Education A+1 (Experimental): Arm: A + 1 Patients received dietary education once. The session focused on phosphorus-rich food identification, dietary restrictions, and basic meal planning.
  Interventions: Behavioral: Nursing education A+1
- Nursing Education A+2 (Experimental): Arm: A + 2 Patients received dietary education twice. The program reinforced dietary knowledge through interactive review and provided individual nutrition tips.
  Interventions: Behavioral: Nursing education A+2
- Nursing Education A+3 (Experimental): Arm: A + 3 Patients received dietary education three times. Sessions included detailed meal planning, food label reading, and repetition to promote long-term adherence.
  Interventions: Behavioral: Nursing education A+3
- Nursing Education B+1 (Experimental): Arm: B + 1 Patients received medication education once. The session introduced phosphate binders, usage timing, and basic instructions for improving adherence.
  Interventions: Behavioral: Nursing education B+1
- Nursing Education B+2 (Experimental): Arm: B + 2 Patients received medication education twice. The intervention emphasized adherence barriers and strategies for taking binders correctly with meals.
  Interventions: Behavioral: Nursing education B+2
- Nursing Education B+3 (Experimental): Arm: B + 3 Patients received medication education three times. The sessions included repeated instruction, practical timing scenarios, and Q&A with nursing staff.
  Interventions: Behavioral: Nursing education B+3
- Nursing Education AB+1 (Experimental): Arm: A+B + 1 Patients received combined dietary and medication education once. The session addressed both phosphorus intake from food and proper medication use.
  Interventions: Behavioral: Nursing education AB+1
- Nursing Education AB+2 (Experimental): Arm: A+B + 2 Patients received combined dietary and medication education twice. The intervention highlighted food-drug interactions and provided dual-domain strategies.
  Interventions: Behavioral: Nursing education AB+2
- Nursing Education AB+3 (Experimental): Arm: A+B + 3 Patients received combined dietary and medication education three times. The sessions offered integrated guidance, practice tools, and individualized plans.
  Interventions: Behavioral: Nursing education AB+3

INTERVENTIONS:
Behavioral: Nursing education A+1 — Dietary education once
  Arms: Nursing Education A+1
Behavioral: Nursing education A+2 — Dietary education twice
  Arms: Nursing Education A+2
Behavioral: Nursing education A+3 — Dietary education three times
  Arms: Nursing Education A+3
Behavioral: Nursing education B+1 — Medication education once
  Arms: Nursing Education B+1
Behavioral: Nursing education B+2 — Medication education twice
  Arms: Nursing Education B+2
Behavioral: Nursing education B+3 — Medication education three times
  Arms: Nursing Education B+3
Behavioral: Nursing education AB+1 — Combined dietary and medication education once
  Arms: Nursing Education AB+1
Behavioral: Nursing education AB+2 — Combined dietary and medication education twice
  Arms: Nursing Education AB+2
Behavioral: Nursing education AB+3 — Combined dietary and medication education three times
  Arms: Nursing Education AB+3

SUMMARY:
By applying statistical methods such as analysis of variance (ANOVA), this study incorporates both the content and the intensity (frequency) of educational interventions to design multiple regression models for evaluating education strategies. Through each round of laboratory data, the investigators aim to identify the most effective educational model using empirical data. The findings will not only improve phosphorus management and enhance the quality of care but also reduce unnecessary nursing workload and help establish an optimal educational protocol and training framework.

Based on literature review and clinical experience, it is well recognized that, in addition to receiving regular and adequate dialysis, effective phosphorus control relies heavily on patients' daily dietary selection and the appropriate use and frequency of phosphate binders. Hence, this study aims to investigate the correlation between phosphorus control and patient education delivered by nursing staff, focusing on dietary management, phosphate binder usage, and knowledge of dialysis principles.

By applying statistical methods such as analysis of variance (ANOVA), this study incorporates both the content and the intensity (frequency) of educational interventions to design multiple regression models for evaluating education strategies. Through each round of laboratory data, we aim to identify the most effective educational model using empirical data. The findings will not only improve phosphorus management and enhance the quality of care but also reduce unnecessary nursing workload and help establish an optimal educational protocol and training framework.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been on dialysis for more than one year, have intact self-awareness, and are currently taking phosphate-binding medications.

Exclusion Criteria:

* Patients who have been on dialysis for less than one year, lack self-awareness, or are not taking phosphate-lowering medications.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
phosphate | Baseline and every 2 weeks until Week 12 (August 19 to November 4, 2025)
  Serum phosphorus levels were measured every two weeks during the 12-week intervention period. Blood samples were collected on Monday or Tuesday, aligned with the patient's hemodialysis cycle (W123 or W246), beginning August 19 and ending November 4, 2025. A total of 6 blood draws were performed. All samples were taken pre-dialysis via venipuncture, with each draw limited to 20 mL and total sample volume not exceeding 320 mL over the study period.
  it is expedited review according to Take blood samples from fingers, heels, ears, or veins of an adult weighing more than 50 kg. Also, the total amount of sample collection should not be more than 320 ml in 8 weeks and should not be more than twice a week. The amount of each blood collection should not be more than 20 ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Wei-Hua, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT07080840/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT07080840/ICF_001.pdf